CLINICAL TRIAL: NCT01967706
Title: A Single-center, Open-label, Randomized, Controlled, Crossover Study to Investigate the Nicotine Pharmacokinetic Profile and Safety of Tobacco Heating System 2.2 Menthol (THS 2.2 Menthol) Following Single Use in Smoking, Healthy Subjects Compared to Menthol Conventional Cigarettes and Nicotine Gum.
Brief Title: Nicotine Pharmacokinetic Profile and Safety of the Tobacco Heating System 2.2 Menthol (THS 2.2 Menthol).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZRHM-PK-05-JP; ZRHM-PK-05-JP (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Smoking
Keywords: Smoking; Nicotine absorption; Candidate modified risk tobacco product; Cigarette; Nicotine replacement therapy; Nicotine gum
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- mTHS then mCC (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of mTHS)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of mCC).
  Interventions: Other: mTHS; Other: mCC
- mCC then mTHS (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of mCC)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of mTHS).
  Interventions: Other: mTHS; Other: mCC
- mTHS then NRT (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single product use of mTHS)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single administration of NRT)
  Interventions: Other: mTHS; Other: NRT
- NRT then mTHS (Active Comparator): Each subject will follow the below study design:
  * Day 0 = Wash-out (1 day)
  * Day 1 = 1st intervention (single administration of NRT)
  * Day 2 = wash-out
  * Day 3 = 2nd intervention (single product use of mTHS).
  Interventions: Other: mTHS; Other: NRT

INTERVENTIONS:
Other: mTHS — Single use of Tobacco Heating System 2.2 Menthol (mTHS)
Other: mCC — Single use of subject's own menthol cigarette (mCC)
  Arms: mCC then mTHS; mTHS then mCC
Other: NRT — Single administration of 2 mg gum (Nicorette® 2mg)
  Arms: NRT then mTHS; mTHS then NRT

SUMMARY:
The primary objective of this clinical study is to evaluate the pharmacokinetic (PK) profile (rate and amount of nicotine absorbed) following a single use of the THS 2.2 Menthol (mTHS), a candidate Modified Risk Tobacco Product, compared to the PK profiles from a single use of a menthol cigarette (mCC) and from a single use of nicotine replacement therapy gum (NRT).

ELIGIBILITY:
Inclusion Criteria:

* Subject is Japanese.
* Smoking, healthy subject as judged by the Investigator.
* Subject has smoked at least 10 commercially available mCCs per day (no brand restrictions) for the last 4 weeks.
* Subject has smoked for at least the last 3 consecutive years.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of a medication (whichever is longer) which has an impact on CYP2A6 activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Fumimasa Nobuoka, MD, Principal Investigator — Ageo Medical Clinic
Locations (1):
- Ageo Medical Clinic, 3133 Haraichi, Ageo-shi, Saitama, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 01 August 2013
  At admission (Day -1), all the subjects performed a product trial (Tobacco Sticks and subsequently NRT gum).
  From enrollment, they were asked to remain abstinent from smoking for at least 24 hours (Day 0) before being randomized on Day 1 into 1 of the 4 sequences.
Pre-assignment Details: Enrolled population = 73 subjects: 11 exposed to mTHS and NRT at Admission but not randomized and 62 randomized as described below:
  * Sequence "mTHS then mCC": 22 subjects
  * Sequence "mCC then mTHS": 22 subjects
  * Sequence "mTHS then NRT": 9 subjects
  * Sequence "NRT then mTHS": 9 subjects
Period: Washout Period of 1 Day (Day 0)
Arm/Group | mTHS Then mCC | mCC Then mTHS | mTHS Then NRT | NRT Then mTHS
Started | 22 | 22 | 9 | 9
Completed | 22 | 22 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: First Intervention (Day 1)
Arm/Group | mTHS Then mCC | mCC Then mTHS | mTHS Then NRT | NRT Then mTHS
Started | 22 | 22 | 9 | 9
Completed | 21 | 22 | 9 | 9
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Washout Period of 1 Day (Day 2)
Arm/Group | mTHS Then mCC | mCC Then mTHS | mTHS Then NRT | NRT Then mTHS
Started | 21 | 22 | 9 | 9
Completed | 21 | 22 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (Day 3)
Arm/Group | mTHS Then mCC | mCC Then mTHS | mTHS Then NRT | NRT Then mTHS
Started | 21 | 22 | 9 | 9
Completed | 21 | 22 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: PK population: all randomized subjects who completed at least 1 of the single-use days, with at least 1 derived PK parameter. Subjects with major protocol deviations impacting the evaluation of the results were excluded.
  62 randomized subjects : 44 in Group 1, 18 in Group 2.
  61 completers: 43 in Group 1 (1 withdrawn subject), 18 in Group 2.
Groups:
- Group 1: This population comprises the following sequences:
  * Sequence "mTHS then mCC"
  * Sequence "mCC then mTHS"
- Group 2: This population comprises the following sequences:
  * Sequence "mTHS then NRT"
  * Sequence "NRT then mTHS"
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 43 | 18 | 61
Age, Customized [Mean (Standard Deviation); unit: years]
  Between 23 and 65 years | 33.4 (10.03) | 30.7 (7.80) | 32.6 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 9 | 29
  Male | 23 | 9 | 32
International Organization for Standardization (ISO) nicotine level [Number; unit: participants]
  ≤ 0.6 mg | 25 | 10 | 35
  > 0.6 to ≤ 1 mg | 18 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) of Nicotine Following Single Use of mTHS, mCC and NRT
Description: T0 = start of single product use.
  Derived from multiple blood sampling on Day 1 and Day 3 (1 blood sampling pre-product use and multiple blood sampling over 24 hours post-product use).
  Geometric Least Squares means are provided.
Time Frame: Blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0
Population: PK populations consisted of all the randomized subjects who completed at least 1 of the single use days (Days 1 or 3), and for whom at least 1 PK parameter could be derived. Subjects with major protocol deviations that impacted the evaluability of the results were excluded from the PK populations.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- mTHS - Group 1; mCC - Group 1: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "mTHS then mCC"
  * Sequence "mCC then mTHS"
- mTHS - Group 2; NRT - Group 2: The geometric least squares mean presented below takes into consideration the data of the subjects who were randomized in the following sequences:
  * Sequence "mTHS then NRT"
  * Sequence "NRT then mTHS"
Arm/Group | mTHS - Group 1 | mCC - Group 1 | mTHS - Group 2 | NRT - Group 2
Number analyzed (Participants) | 43 | 43 | 18 | 18
ng/mL | 10.70 [8.94 to 12.80] | 12.09 [10.10 to 14.47] | 7.64 [5.39 to 10.81] | 7.52 [5.31 to 10.64]
Statistical Analysis 1: Comparison: mTHS - Group 1 vs mCC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of mTHS:mCC) for Cmax, therefore, there was no statistical hypothesis to be tested for this objective; Test type: Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 88.47, 95% CI 2-sided [68.64 to 114.03] — LS mean ratio (mTHS - Group 1:mCC - Group 1)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (Pre-product Use) to Last Time Point [AUC(0-last)] Following Single Use of mTHS, mCC and NRT
Description: as for outcome 1
Time Frame: Blood taken 15 minutes prior to T0, 2, 4, 6, 8, 10, 15, 30, 45 minutes, 1, 2, 4, 6, 9, 12, and 24 hours after T0
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | mTHS - Group 1 | mCC - Group 1 | mTHS - Group 2 | NRT - Group 2
Number analyzed (Participants) | 43 | 43 | 18 | 18
ng*h/mL | 23.99 [20.87 to 27.57] | 24.45 [21.27 to 28.10] | 15.61 [11.96 to 20.37] | 27.94 [21.41 to 36.45]
Statistical Analysis 1: Comparison: mTHS - Group 1 vs mCC - Group 1; The objective of this study was to determine the point estimate and precision of the nicotine bioavailability (ratio of mTHS:mCC) for AUC(0-last), therefore, there was no statistical hypothesis to be tested for this objective; Test type: Other; ANOVA; The model included terms for sequence, subject nested within sequence, period, and product as fixed effect factors; Geometric LS Mean Ratio = 98.13, 95% CI 2-sided [80.61 to 119.46] — LS mean ratio (mTHS - Group 1:mCC - Group 1)

ADVERSE EVENTS:
Time Frame: From informed consent form (ICF) signature until the end of the safety follow-up period (7 days after discharge of the subject).
Description: The safety was assessed in the safety population, consisting of 73 subjects: 62 randomized subjects (44 in Group 1, 18 in Group 2) and 11 subjects exposed to mTHS and NRT from the product trials on Day -1 but not randomized.
Groups:
- Group 1: This population comprised the subjects that followed these intervention sequences:
  * Sequence "mTHS then mCC"
  * Sequence "mCC then mTHS"
- Group 2: This population comprised the subjects that followed these intervention sequences:
  * Sequence "mTHS then NRT"
  * Sequence "NRT then mTHS"
- Enrolled But Not Randomized: Subjects who tried the mTHS at Admission (Day -1) but were not randomized in 1 of the 2 groups as they were back-up subjects
Arm/Group | Group 1 | Group 2 | Enrolled But Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 0/44 | 1/18 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=44) | Group 2 (N=18) | Enrolled But Not Randomized (N=11)
Hemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2013-06-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT01967706/Prot_000.pdf
  • Statistical Analysis Plan (2014-05-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT01967706/SAP_001.pdf